CLINICAL TRIAL: NCT06327763
Title: Prophylactic Ilioinguinal Neurectomy During Open Tension-Free Inguinal Hernia Repair for Prevention of Chronic Postoperative Pain
Brief Title: Prophylactic Ilioinguinal Neurectomy During Open Tension-Free Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Yasser Ali Orban, assisstant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ilioinguinal Neurectomy
Record Dates: First submitted 2024-03-16; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Ilioinguinal Nerve Section; Pain Prevention; Hernioplasty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inguinal hernioplasty with ilioinguinal nerve preservation (No Intervention)
- inguinal hernioplasty with ilioinguinal nerve section (Experimental)
  Interventions: Procedure: ilioinguinal nerve section

INTERVENTIONS:
Procedure: ilioinguinal nerve section — patients operated on by open inguinal hernioplasty with ilioinguinal neurectomy
  Arms: inguinal hernioplasty with ilioinguinal nerve section

SUMMARY:
postoperative chronic inguinal pain is a common postoperative complication after open inguinal hernia repair.

Chronic inguinal pain is a common complication following open inguinal hernia repair. Ilioinguinal nerve entrapment is a common cause of this chronic pain which may adversely affect the patients' life. Ilioinguinal neurectomy seems to be beneficial in preventing such pain, but it carries the risk for numbness and hypoesthesia.

ELIGIBILITY:
Inclusion Criteria:

- the study included all adult patients operated on for unilateral inguinal hernia by Lichtenstein tension-free mesh hernioplasty with or without ilioinguinal neurectomy.

Exclusion Criteria:

* patients with recurrent inguinal hernia, bilateral inguinal hernia repair, or huge inguinoscrotal hernia were excluded. Diabetic patients as well as, patients with suspected inguinal hernia recurrence at the time of the questionnaire were excluded.

Ages: 16 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 196 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
detect postoperative pain using short form inguinal pain questionnaire | 3 months following operation then continous
  ask the patient for presence of postoperative pain using short form inguinal pain questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- yasmine Hegab, Zagazig, Egypt

REFERENCES:
- [Derived] Orban YA, Hegab YH, Hamed AEM, Metwally H, Zakaria R, Goda AM, Baz Y. Prophylactic triple neurectomy during open tension-free inguinal hernia repair: a clinical trial for the prevention of chronic postoperative pain. Updates Surg. 2026 Jan 22. doi: 10.1007/s13304-025-02497-3. Online ahead of print. PMID 41571965